CLINICAL TRIAL: NCT02316522
Title: Epigenetic Contribution to the Pathogenesis of Diabetic Nephropathy in Qatari Population
Status: Completed | Type: Observational
Sponsor: Weill Medical College of Cornell University (Other)
Collaborators: Hamad Medical Corporation (Industry); Weill Cornell Medical College in Qatar (Other)
Responsible Party: Sponsor
Other Study IDs: 14-00043 [JIRB]
Record Dates: First submitted 2014-12-09; First posted 2014-12-15 (Estimated); Last update posted 2022-05-02 (Actual); Status verified 2022-04

CONDITIONS: Type 2 Diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood Urine
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (4):
- Group I: T2D nephropathy: Individuals with type 2 diabetes and nephropathy
- Group II: T2D and no nephropathy: Individuals with type 2 diabetes and no nephropathy
- Group III: Control, non-diabetic: Non-diabetic individuals with normal kidney function
- Group IV: Controls, non-diabetic: Non-diabetic individuals with hypertensive nephropathy

SUMMARY:
The main objective is to study the epigenetic contribution to the pathophysiology of diabetic nephropathy in Qatari population.

DETAILED DESCRIPTION:
Diabetic nephropathy (DN) is a common vascular complication of Type 2 diabetes (T2D) that is associated with increased mortality and poor quality of life.In industrialized countries, DN ranges first among other etiologies of end-stage renal disease (ESRD).Diabetes in Qatar is a serious health issue for the Qatari population since approximately 1/5 of the population has T2D, which is 2-3 times higher than the world average. As observed in other Gulf cooperation council (GCC) countries, obesity and sedentary lifestyle are cornerstones in the development of T2D. Additionally, consanguineous marriages in Qatar contribute to this high prevalence. As a consequence, DN has an enormous burden in terms of management, treatment and especially in renal replacement therapy (RRT) in ESRD in Qatari Population.DN is a glomerular disease defined by increased urinary albumin excretion (UAE), hypertension and decline in the glomerular filtration rate (GFR), all induced by chronic hyperglycemia. However, there are other contributing factors such as genetic predisposition, systemic and intra-renal hemodynamic disturbances, all leading to glomerulosclerosis. All of the known pathways do not explain the complex pathophysiology behind DN. Even different variants of genes described in major GWAS studies have little impact in terms of risk prevention or prognosis of DN. Over the last decade, epigenetics have initiated a new era in Genetic Medicine capable of giving a different approach to human disease.

ELIGIBILITY:
Inclusion Criteria:

* Males and females, at least 18 years old
* Provide informed consent
* Willingness to participate in the study
* In patients with diabetes, no concomitant diseases except for micro and macrovascular complications of diabetes (nephropathy, retinopathy, peripheral arterial disease, coronary artery disease, neuropathy) or symptoms of the metabolic syndrome ( hypertension, dyslipidemia and obesity)
* Not taking any chronic medications (except of the diabetes and the cardiovascular related drugs)
* Consent to having peripheral blood and urine collection for DNA extraction and micro-RNAs as well as routine laboratory evaluation, including general hematologic studies, general biochemical analyses.

Exclusion Criteria:

* Type I diabetes or other form of diabetes (MODY, secondary diabetes)
* Unable to meet the inclusion criteria
* Pregnancy
* Active infection or acute illness of any kind
* Chronic inflammation (auto-immune diseases) or infections (HIV, chronic viral hepatitis, chronic urinary tract infections …)
* Evidence of malignancy within the past 5 years
* Chronic hematological disorders known to affect glycated hemoglobin results such as hemoglobinopathies and pathologies with high red-cell turnover

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Subjects will be recruited from Hamad Medical Corporation.
Sampling Method: Non-Probability Sample
Enrollment: 158 (Actual)
Dates: Start 2014-10-23 (Actual); Primary Completion 2018-04-09 (Actual); Study Completion 2018-04-09 (Actual)

PRIMARY OUTCOMES:
DNA methylation | 1 hr
  Assess DNA methylation in monocytes

SECONDARY OUTCOMES:
Micro-RNAs | 1 hr
  Assess urinary micro-RNAs

CONTACTS AND LOCATIONS:
Overall Officials: Charbel Abi Khalil, MD, Principal Investigator — Weill Cornell Medical College in Qatar
Locations (1):
- Hamad Medical Corporation, Doha, Qatar

IPD SHARING:
Plan to Share IPD: Undecided